CLINICAL TRIAL: NCT02114112
Title: Randomised Controlled Trial to Study the Effect of Nasal Continuous Positive Airway Pressure (NCPAP) Cycling on Successful Weaning When Compared With Nasal Continuous Positive Airway Pressure (NCPAP) in Premature Infants of 25-28 Weeks Gestation
Brief Title: E-23596 - Use of NCPAP Cycling to Wean Preterm Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to new respiratory quality control initiative introduced in the NICU, recruitment for the study was stopped.
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, ABHAY LODHA, Staff Neonatologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-23596
Record Dates: First submitted 2014-04-06; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Premature Birth
Keywords: Bronchopulmonary dysplasia; Continuous positive airway pressure pressure; Preterms
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A-NCPAP Cycling group (Experimental): Infants in Group A were cycled between NCPAP and nasal prongs. For the first 12 hours, infants received 10 hours of NCPAP and 2 hours of 1 litre per minute of nasal prongs (NP). For the next 12 hours, infants received 8 hours of NCPAP and 4 hours of NP. In the subsequent 24 hours, infants alternated between 6 hours of NCPAP and 6 hours of NP. In the last 24 hours of intervention they alternated between 4 hours of NCPAP and 8 hours of NP.
  Interventions: Other: NCPAP cycling
- Group B-Continuous NCPAP (Active Comparator): Infants randomized to group B received continuous NCPAP at a CPAP distending pressure of 4 cm of water for 72 hours. Both the groups after 72 hours of intervention were weaned to 1litre per minute NP. During the intervention period all infants were scored using the ACoRN respiratory score on a 12 hourly basis.
  Interventions: Other: NCPAP continuous

INTERVENTIONS:
Other: NCPAP cycling
  Arms: Group A-NCPAP Cycling group
Other: NCPAP continuous
  Arms: Group B-Continuous NCPAP

SUMMARY:
Objective: To compare the effectiveness of nasal continuous positive airway pressure (NCPAP) cycling to continuous NCPAP in successful weaning of preterm infants of 25-28 weeks gestation to nasal prongs.

Methods: A total of 40 infants with a gestational age (GA) of 25-28 weeks ventilated for respiratory distress syndrome (RDS) and extubated to NCPAP are eligible for the study. They will be randomized to NCPAP cycling {Group A; cycling between NCPAP of 4 cm and 1litre per minute of nasal prongs} or to continuous CPAP at 4 cm of water (Group B). Primary outcome is the number of babies who came off NCPAP at the end of 72 hours of the intervention and remained off NCPAP for the next 72 hours. The duration of NCPAP, Bronchopulmonary dysplasia (BPD) at 36 weeks post menstrual age and Retinopathy of Prematurity (ROP) stage ≥3 will be the secondary outcomes.

DETAILED DESCRIPTION:
Randomized Controlled Trial to Study the Effect of Nasal Continuous Positive Airway Pressure (NCPAP) Cycling on Successful Weaning when Compared with Continuous Nasal Positive Airway Pressure (NCPAP) in Premature Infants of 25-28 weeks gestations Background: In Canada, preterm babies of < 28 weeks gestation constitute 12% of all newborn admissions and their survival has increased from 65% to 72%. In Alberta, the premature birth rate has been increasing over the past several years and although these preterm infants make up a small percentage of births, they add disproportionately to the mortality, morbidity and cost of medical care. Their rate of long-term neurodevelopmental disability is also disproportionately high. Advances in neonatal ventilation and neonatal care including increased use of antenatal steroids, postnatal surfactant, improved mechanical ventilation and early use of total parenteral nutrition have improved survival of extremely low birth weight (ELBW) premature infants. Despite these advances, the incidence of Bronchopulmonary Dysplasia (BPD) in these infants remains high in Southern Alberta.

Perinatal risk factors and the duration of mechanical ventilation, including high inspired oxygen, high peak inspiratory pressure, lower positive end-expiratory pressure, higher ventilation rate and hypocarbia (Partial pressure of carbon dioxide < 40 cm of water at 48 to 96 hours) are associated with later development of BPD in these premature infants. Although pressure-induced injury might play a role in the injury leading to 'new' BPD, alveolar over distention is likely to be a more important contributing factor. Atelectasis also contributes to BPD as ventilation of the atelectatic lung leads to pulmonary parenchymal injury through the sheer stress of repeatedly reinflating collapsed alveoli. Despite various preventive and treatment strategies including permissive hypercapnia, high frequency ventilation, antioxidants, indomethacin, fluid restriction and use of diuretic, the prevalence of BPD continues to be unacceptably high. It is unclear whether minimum ventilator pressure exposure to premature lungs could prevent increasing incidence of BPD with the use of nasal continuous positive airways pressure (NCPAP) cycling ( NCPAP for a few hours alternating with continuous nasal flow) when compared with continuous NCPAP. High pressure on the ventilator or continuous NCPAP possibly remains an underlying mechanism for pressure and volume induced injury to the lungs and exhaustion of the respiratory muscle.

Prolonged ventilation may predispose diaphragmatic myofibrils to disuse atrophy or failure of normal growth, which contributes, to difficulties in weaning infants from mechanical ventilator support including Nasal continuous positive airways pressure (NCPAP). Age and gestation dependent changes in contractile function of the diaphragm include decreased fatigue resistance with advancing maturation and Ventilator Induced Diaphragmatic Dysfunction (VIDD). The combination of high work, rapid breathing, and low-oxidative capacity suggests respiratory muscle fatigue in the infant with respiratory disease. Even short-term controlled mechanical ventilation produces significant remodeling and functional alterations of the diaphragm, which could impede efforts at discontinuing ventilator support.

Prolonged use of mechanical ventilation has also been associated with infections, subglottic stenosis and aspiration. Therefore, clinicians strive to wean early from the ventilator and avoid reintubation once infants are extubated. Clinical signs of respiratory failure after extubation include apnea (prolonged cessation of respiration for 20 seconds or more and/or associated with cyanosis; abrupt, marked pallor or hypotonia; bradycardia), respiratory acidosis or increasing oxygen requirements. These problems may lead to reintubation and ventilation with their attendant morbidity and economic costs. NCPAP appears to stabilize the upper airway, improve lung function and reduce apnea. Randomized trials have shown that NCPAP, applied prophylactically after extubation, reduces the need for additional ventilatory support and is associated with a lower incidence of BPD compared to mechanical ventilation. NCPAP supports the compliant chest wall of the neonate by providing a pneumatic splint to counteract the tendency to move paradoxically during inspiration or to collapse upon expiration. NCPAP has been used to prevent extubation failure and as an alternative to intubation and ventilation for respiratory distress syndrome in very preterm infants. The optimal method of weaning infants from NCPAP remains unanswered. Although some Neonatal intensive care units try abrupt discontinuation of NCPAP, most wean on an ad hoc basis by gradually decreasing either time spent on the Infant Flow Driver (IFD) or the NCPAP pressure. Early discontinuation of NCPAP may carry the risk of pulmonary atelectasis, apnea and bradycardia. The most common reason for failure to wean on NCPAP is respiratory acidosis, apneas, bradycardias, and increasing oxygen requirements above 60%. Similarly, the most common reason for re-ventilation is respiratory acidosis. In a prospective study in 2011 on preterm infants with resolving respiratory distress syndrome, NCPAP impeded systemic and pulmonary venous return but did not compromise systemic arterial pressure or heart rate. The important issue, therefore, is the rationale of continuing NCPAP when supplemental oxygen requirement have ended, in the absence of moderate-to-severe apnea. Mechanical ventilation and NCPAP both tend to cause barotraumas and possibly BPD in premature infants. It is unclear whether preterm infants who undergo NCPAP cycling with free flow of oxygen are at less risk for BPD compared to those who are dependent on continuous NCPAP. In a randomized controlled trial of discontinuation of NCPAP in 2011, authors found that almost all preterm infants breathing room air tolerated a 6 hour pause in NCPAP with no increase in apnea and bradycardia. A reduction in the subsequent use of NCPAP was also observed. These findings led to the development of a strategy to further reduce ventilator induced trauma and thus BPD. This strategy used non-invasive intermittent continuous positive airway pressure ventilation by alternating NCPAP with continuous nasal flow (CNF) via nasal prongs for ELBW infants. This method of ventilation is termed cycling of NCPAP. In our subjective clinical experience, cycling of NCPAP with CNF reduces the duration of respiratory support and therefore would be expected to reduce the incidence of BPD. Cycling reduces duration of NCPAP and dependency, trauma and or deviation of nasal septum, feed intolerance due to gastric distension, agitation from pain/discomfort and nosocomial infection. The benefits of cycling NCPAP in comparison to continuous NCPAP in premature infants have not been studied in clinical trials. The aim of this pilot study is to establish the ability of NCPAP cycling to prevent reintubation, decrease the duration of respiratory support and thereby, the incidence of BPD.

Rationale for this study: There is no evidence in the literature that premature infants who are treated with NCPAP cycling alternating with continuous nasal air flow (CNF) versus NCPAP without alternating CNF do better or worse in the immediate newborn period. We speculate that NCPAP cycling or weaning will gradually shift the work of breathing from the supportive intervention to the baby without producing fatigue of respiratory muscles and trauma to the developing lungs. Currently, this mode of respiratory support is being used in our Neonatal intensive care unit. It is largely determined by personal preferences with little clinical data, only experimental or anecdotal evidence without any long-term outcomes data. A retrospective study to confirm benefits of cycling NCPAP with CNF versus continuous NCPAP is not feasible since duration of this alternative therapy has varied in infants of different gestational ages. There is equipoise regarding the role of cycling NCPAP with CNF versus continuous NCPAP without CNF in premature infants. Therefore, it would be prudent to study the benefits of NCPAP cycling versus continuous NCPAP in premature infants. Our pilot study will address the importance of NCPAP cycling as a useful weaning mode in ELBW infants. Results of this pilot study will inform future power and sample size calculations for a larger randomized controlled trial. Information obtained from this study will also fill gaps in the existing knowledge in neonatal medicine and will resolve current controversies concerning the use of NCPAP cycling with CNF versus continuous NCPAP in ELBW infants.

Hypothesis: We hypothesize that more infants receiving NCPAP cycling with CNF will successfully wean to nasal prongs in 72 hours compared with continuous NCPAP.

Rationale for pilot study: Our pilot study is an initial or preliminary investigation designed to test research hypothesis, gather data, and validate the scientific approach and methodology for NCPAP with CNF cycling versus continuous NCPAP. Results of this study will be an applied to designing a randomized controlled trial and in applying for an operating grant.

Research Question: Does the use of NCPAP cycling with CNF in preterm infants of 25-28 weeks gestation enable successful weaning of babies to nasal prongs in 72 hours when compared to continuous NCPAP?

Objective: The purpose of this study is to determine if a regimen on NCPAP with CNF will be more successful in weaning babies to nasal prongs in 72 hours compared with continuous NCPAP in premature infants.

Research Methods: 1. Study Design: We propose a prospective, open label, pilot, randomized controlled trial of two different methods of respiratory support after extubation in premature infants in Neonatal intensive care unit. The two methods of respiratory supports are alternating NCPAP and CNF versus continuous NCPAP.

2. Subjects specifications: Settings: The study will be conducted in the level III Neonatal intensive care unit at the Foothills Medical Centre in Calgary, Alberta.

Target population: All premature infants 25-28 weeks gestational age admitted to Neonatal intensive care unit.

Sample selection: Infants will be identified according to inclusion and exclusion criteria (described below). After obtaining informed consent from their parent(s), they will be randomized and included in the study.

3.Randomization: This will be achieved using a computerized random number generator. We will use random block sizes of 2 and 4 to increase the likelihood of equal enrolment into each group. Randomization procedure will occur on site, will be concealed and undertaken by health personnel who will be not involved in our study. Treatment allocation cards will be wrapped in foil and inserted into opaque sequentially numbered sealed envelopes which will be kept in a locked drawer in the Neonatal intensive care unit. Envelopes will be opened sequentially at the time of allocation. 4. Inclusion criteria: All premature infants born between 25-28 weeks gestation, ventilated for respiratory distress syndrome (RDS) and extubated to NCPAP for at least 72hours are eligible. RDS will be defined by clinical criteria and radiological findings. 5. Exclusion criteria: Infants with major congenital anomalies including complex heart disease, central causes for respiratory depression, persistent pulmonary hypertension and air leaks will be excluded from the study. 6. Recruitment: Infants meeting the inclusion/exclusion criteria were identified and investigators approached their parents during the early clinical course while the baby is still ventilated to obtain informed written consent.

7. Intervention: Predefined extubation criteria were used in guiding the decision to extubate infants. The criteria for extubation are peak inspiratory pressure of 16 cm water, positive end expiratory pressure of 5 cm of water, intermittent mandatory ventilation rate of 10 to 20 and fraction of inspired oxygen 0.30 or based on attending physician's decision. Two hours prior to extubation, infants were started on caffeine therapy. All infants were extubated to Infant Flow Driver NCPAP as per standard practice. Infants, who remain on NCPAP for at least 72 hours and meet the Weaning from NCPAP criteria, were randomized to either the Weaning regimen with cycling or the continuous NCPAP regimen without cycling.

Weaning regimen in intervention arm: The weaning protocol was as follows:- 10 hours on NCPAP followed by 2 hours on binasal Hudson's nasal cannula at 1litre per minute flow for 12 hours 8 hours on NCPAP followed by 4 hours on binasal Hudson's nasal cannula at 1litre per minute flow for 12 hours 6 hours on NCPAP followed by 6 hours on binasal Hudson's nasal cannula at 1litre per minute flow for 24 hours 4 hours on NCPAP followed by 8 hours on binasal Hudson's nasal cannula at 1litre per minute flow for 24 hours Each infant was assessed following every 12-hour period clinically, with blood gases and a chest radiograph at the end of the first cycle & at the end of intervention. Continuous NCPAP regimen: After the infant is randomized to this group, he/she was placed on Infant Flow Driver CPAP at a pressure of 4 cm of water for 72 hours continuously. At the end of 72 hours, the infant was weaned to NP at 1litre per minute. If an infant meets the failure criteria, continuous NCPAP was restarted. Blood gas analysis was done at 12-hour intervals, which is in keeping with the standard of care for monitoring infants who are being weaned off of respiratory support. The infant's ACoRN score will be plotted every 12 hours or sooner if there is an acute deterioration. Success was defined as remaining off NCPAP for 72hours after the intervention. Weaning from NCPAP Criteria: 1) ACoRN respiratory score≤4 and 2) NCPAP pressures equal to 5 cm of water and 3) Supplemental oxygen requirement less than 40% and 4) potential of hydrogen (pH) >7.25 and 5) Tolerating time off NCPAP well during nursing care.

Failure Criteria:

1. ACoRN respiratory score ≥5 or increase from previous score by 2 points in a 12 hour period or
2. supplemental oxygen more than 50% or
3. acidosis with pH<7.25 or
4. apnea with bradycardia or desaturation requiring stimulation >1/hour or
5. apneic episode requiring Positive Pressure Ventilation with Bag & Mask in a 12 hour period. Criteria to Reintubate at any point during the study include

1) Acidosis with pH ≤7.2 or two consecutive pH≤7.25 or 2) Fractional inspired oxygen more than 50% or Partial pressure of carbon dioxide ≥70 or 3) Severe recurrent apnea (≥2 apneas requiring intermittent positive-pressure ventilation).

Oxygen concentration will be titrated by the clinical team to achieve a transcutaneous oxygen saturation of between 88 and 92% as per the policy in our neonatal intensive care unit.

Data collection:

Primary Outcome: Number of babies who came off the NCPAP at the end of 72 hours of the intervention and remained off NCPAP for 72 hours.

Secondary Outcome:

1. Total duration of NCPAP after the intervention,
2. BPD at 36 weeks of post-conceptional age,
3. ROP stage 3 and more Additional data collection: gestational age, birth weight, RDS, antenatal steroids, surfactant treatment, sepsis, Intraventricular hemorrhage, Patent ductus arterioses, pneumonia, pulmonary hemorrhage, Necrotizing enterocolitis. A data collection form will be used to gather information regarding the antenatal history, birth data, and details of ventilation, details of intervention, complications and outcome.

Statistical considerations Sample size: Since this was a pilot study the investigators planned to enroll 20 premature infants in each group by randomization. The results of this study will help to plan a complete randomized controlled trial. For full study sample size estimation: The sample size estimates will be based on the results obtained from our pilot study.

Data analysis: Data was analyzed using statistical package statistical analysis system (SAS) with the assistance of a biostatistician. A test for difference in proportions was performed and a 95% confidence interval for the difference provided. Student's t-test was used for continuous variables where the data is normally distributed and Chi square-test for categorical data.

Ethical Considerations: The study was submitted to the research ethics board of University of Calgary. Confidentiality of patient data was enforced throughout the study. Study number identified each patient only. Written informed consent was obtained from parents prior to enrolment in the study. Participation in the study was voluntary and parents were allowed to withdraw their infants at any time during the study period.

Feasibility of the study: In the year 2009, a total of 110 infants were born between 25 and 28 weeks gestation at Foothills Medical Centre. Therefore investigators planned to complete the study within two years.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 25-28 weeks gestation
* Ventilated for respiratory distress syndrome (RDS)
* Extubated to NCPAP for at least 72 hours.

Exclusion Criteria:

* Major congenital
* Chromosomal anomalies.

Ages: 72 Hours to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Successful weaning off NCPAP at the end of 72 hours of the intervention. | 72 hours
  Primary outcome was successful weaning off NCPAP at the end of 72 hours of the intervention and remained off NCPAP for the next 72 hours

SECONDARY OUTCOMES:
The duration of NCPAP | 36 weeks post menstrual age
Bronchopulmonary dysplasia | 36 weeks post mentstrual age
Retinopathy of prematurity stage 3 or higher | 36 weeks post menstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Lodha, MD, DM,MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Room C211, 1403 - 29th Street NW, Calgary, Alberta, Canada